CLINICAL TRIAL: NCT04829370
Title: Clinical Application of Patented Lyophilized PLT in Acne Scar Repairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Collaborators: Spirit Scientific (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20170903R
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Atrophic Acne Scar
Keywords: Platelet; PLT; Growth factor; Acne scar repairment; Laser
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A prospective, single-blind, parallel study at a single health care center.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLT (Active Comparator): All subjects are treated with fractional carbon dioxide laser, then applied 2 mL PLT solution (dissolved in normal saline) on the right face.
  Interventions: Other: PLT
- Saline (Placebo Comparator): All subjects are treated with fractional carbon dioxide laser, the left face (control group) be applied 2 mL normal saline
  Interventions: Other: Saline

INTERVENTIONS:
Other: PLT — The study will be conducted by using a fractional carbon dioxide laser for acne scar treatment. After the treatment, each patient enrolled will be applied 2 mL PLT solution on the right face. Treatment mentioned above will be repeated every 3 to 4 weeks, overall 4 times treatment and one month follow up after fourth treatment. Every record will be documented in questionnaires by the principal investigator and the patient itself. Moreover, VISIA is applied for objective observation, such as spots, wrinkles, texture, pores, UV spots, brown spots, red area, and porphyrins could be objectively analyzed.
  Arms: PLT
Other: Saline — The study will be conducted by using a fractional carbon dioxide laser for acne scar treatment. After the treatment, each patient enrolled left face be applied 2 mL normal saline.
  Treatment mentioned above will be repeated every 3 to 4 weeks, overall 4 times treatment and one month follow up after fourth treatment. Every record will be documented in questionnaires by the principal investigator and the patient itself. Moreover, VISIA is applied for objective observation, such as spots, wrinkles, texture, pores, UV spots, brown spots, red area, and porphyrins could be objectively analyzed.
  Arms: Saline

SUMMARY:
All kinds of skin problems will cause a person's life caused by varying degrees of trouble, especially issues at face. No matter diseases or aging would cause mental pressure and the inconvenience in different ages.

Scar caused by acne is the most common skin issue amount young people. While acne recovering, due to the destruction of collagen forming fibrous tissue, and scars be left. Clinical treatments are facial laser, argon laser and carbon dioxide laser. With the combination of rejuvenation to accelerate growth of collagen when needed. According to journal articles, facial laser combined with Platelet-rich plasma is more curative than facial laser treatment alone and can significantly reduce side effects (Dermatol Surg. 2014 Feb;40(2):152-61).

Platelet has been valued in regeneration medicine due to its various growth factors with repairment, induction and promotion functions. Moreover, low risk of allergy for it is an autologous material. Platelet had been officially applied in orthopedics and more clinical studies in many other fields. Nowadays, preparation of PRP is by single-use centrifuge tube, patients have to go through blood collection process every time before therapy due to short shelf life of PRP. Meanwhile, amount of platelet in PRP would be different due to difference of individual, health condition and separation methods. Thus, leaving unknown of active principle and uncertainty of treatments.

In this trial, a patented technique of lyophilized PLT preparation method is applied, collect 250 c.c. of blood specimen by using blood bag, separate platelet in germ-free clean room, then lyophilize platelet to extend shelf life to at least three years after quantifying platelet amount. Therefore, treatment could be done after simple dissolution process of PLT leads to the convenience of multiple therapy lessons.

ELIGIBILITY:
Inclusion Criteria:

- all subjects of acne scars are defined of grades 1, 2, and 3 [Goodman and Baron Grading scale] were enrolled in the study.

Exclusion Criteria:

* Exclusion criteria included treatment with any laser device treatment to the face within 1 month, use of systemic retinoids within 3 months, pregnancy or lactation, a history of hypertrophic scarring or keloids, cancer therapies, uncontrolled diabetes, chronic liver or kidney disease, cardiovascular disease or hematologic disorders. Subjects were requested to avoid using any topical products containing alpha-hydroxy acids and salicylic acid on the face during the study period.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
adverse effect assessment | 20 weeks
  adverse effect assessment, Safety

SECONDARY OUTCOMES:
Global assessment of acne scar | 20 weeks
  5-point grading of acne scar
wound healing rate | 20 weeks
  7-days grading of wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Chieh-Chen Huang, Shin Kong Wu Ho Su Memorial, M, Principal Investigator — Department of Dermatology, Shin Kong Wu Ho Su Memorial Hospital,
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Ghodsi SZ, Orawa H, Zouboulis CC. Prevalence, severity, and severity risk factors of acne in high school pupils: a community-based study. J Invest Dermatol. 2009 Sep;129(9):2136-41. doi: 10.1038/jid.2009.47. Epub 2009 Mar 12. PMID 19282841
- [Background] Collier CN, Harper JC, Cafardi JA, Cantrell WC, Wang W, Foster KW, Elewski BE. The prevalence of acne in adults 20 years and older. J Am Acad Dermatol. 2008 Jan;58(1):56-9. doi: 10.1016/j.jaad.2007.06.045. Epub 2007 Oct 22. PMID 17945383
- [Background] Layton AM. Optimal management of acne to prevent scarring and psychological sequelae. Am J Clin Dermatol. 2001;2(3):135-41. doi: 10.2165/00128071-200102030-00002. PMID 11705090
- [Background] Moradi Tuchayi S, Makrantonaki E, Ganceviciene R, Dessinioti C, Feldman SR, Zouboulis CC. Acne vulgaris. Nat Rev Dis Primers. 2015 Sep 17;1:15029. doi: 10.1038/nrdp.2015.29. PMID 27189872
- [Background] Connolly D, Vu HL, Mariwalla K, Saedi N. Acne Scarring-Pathogenesis, Evaluation, and Treatment Options. J Clin Aesthet Dermatol. 2017 Sep;10(9):12-23. Epub 2017 Sep 1. PMID 29344322
- [Background] Fabbrocini G, Annunziata MC, D'Arco V, De Vita V, Lodi G, Mauriello MC, Pastore F, Monfrecola G. Acne scars: pathogenesis, classification and treatment. Dermatol Res Pract. 2010;2010:893080. doi: 10.1155/2010/893080. Epub 2010 Oct 14. PMID 20981308
- [Background] Dunn LK, O'Neill JL, Feldman SR. Acne in adolescents: quality of life, self-esteem, mood, and psychological disorders. Dermatol Online J. 2011 Jan 15;17(1):1. PMID 21272492
- [Background] Sanchez Viera M. Management of acne scars: fulfilling our duty of care for patients. Br J Dermatol. 2015 Jul;172 Suppl 1:47-51. doi: 10.1111/bjd.13650. PMID 25597636
- [Background] Ong MW, Bashir SJ. Fractional laser resurfacing for acne scars: a review. Br J Dermatol. 2012 Jun;166(6):1160-9. doi: 10.1111/j.1365-2133.2012.10870.x. Epub 2012 May 8. PMID 22296284
- [Background] Manuskiatti W, Triwongwaranat D, Varothai S, Eimpunth S, Wanitphakdeedecha R. Efficacy and safety of a carbon-dioxide ablative fractional resurfacing device for treatment of atrophic acne scars in Asians. J Am Acad Dermatol. 2010 Aug;63(2):274-83. doi: 10.1016/j.jaad.2009.08.051. PMID 20633798
- [Background] Sclafani AP, Romo T 3rd, Ukrainsky G, McCormick SA, Litner J, Kevy SV, Jacobson MS. Modulation of wound response and soft tissue ingrowth in synthetic and allogeneic implants with platelet concentrate. Arch Facial Plast Surg. 2005 May-Jun;7(3):163-9. doi: 10.1001/archfaci.7.3.163. PMID 15897404
- [Background] Hom DB, Linzie BM, Huang TC. The healing effects of autologous platelet gel on acute human skin wounds. Arch Facial Plast Surg. 2007 May-Jun;9(3):174-83. doi: 10.1001/archfaci.9.3.174. PMID 17519207
- [Background] Dougherty EJ. An evidence-based model comparing the cost-effectiveness of platelet-rich plasma gel to alternative therapies for patients with nonhealing diabetic foot ulcers. Adv Skin Wound Care. 2008 Dec;21(12):568-75. doi: 10.1097/01.ASW.0000323589.27605.71. PMID 19065083
- [Background] Jee CH, Eom NY, Jang HM, Jung HW, Choi ES, Won JH, Hong IH, Kang BT, Jeong DW, Jung DI. Effect of autologous platelet-rich plasma application on cutaneous wound healing in dogs. J Vet Sci. 2016 Mar;17(1):79-87. doi: 10.4142/jvs.2016.17.1.79. Epub 2016 Mar 22. PMID 27051343
- [Background] Tambella AM, Attili AR, Dupre G, Cantalamessa A, Martin S, Cuteri V, Marcazzan S, Del Fabbro M. Platelet-rich plasma to treat experimentally-induced skin wounds in animals: A systematic review and meta-analysis. PLoS One. 2018 Jan 11;13(1):e0191093. doi: 10.1371/journal.pone.0191093. eCollection 2018. PMID 29324848
- [Background] Leo MS, Kumar AS, Kirit R, Konathan R, Sivamani RK. Systematic review of the use of platelet-rich plasma in aesthetic dermatology. J Cosmet Dermatol. 2015 Dec;14(4):315-23. doi: 10.1111/jocd.12167. Epub 2015 Jul 23. PMID 26205133
- [Background] Shin MK, Lee JH, Lee SJ, Kim NI. Platelet-rich plasma combined with fractional laser therapy for skin rejuvenation. Dermatol Surg. 2012 Apr;38(4):623-30. doi: 10.1111/j.1524-4725.2011.02280.x. Epub 2012 Jan 30. PMID 22288389
- [Background] Zhu JT, Xuan M, Zhang YN, Liu HW, Cai JH, Wu YH, Xiang XF, Shan GQ, Cheng B. The efficacy of autologous platelet-rich plasma combined with erbium fractional laser therapy for facial acne scars or acne. Mol Med Rep. 2013 Jul;8(1):233-7. doi: 10.3892/mmr.2013.1455. Epub 2013 May 2. PMID 23653117
- [Background] Gawdat HI, Hegazy RA, Fawzy MM, Fathy M. Autologous platelet rich plasma: topical versus intradermal after fractional ablative carbon dioxide laser treatment of atrophic acne scars. Dermatol Surg. 2014 Feb;40(2):152-61. doi: 10.1111/dsu.12392. Epub 2013 Dec 19. PMID 24354616
- [Background] Na JI, Choi JW, Choi HR, Jeong JB, Park KC, Youn SW, Huh CH. Rapid healing and reduced erythema after ablative fractional carbon dioxide laser resurfacing combined with the application of autologous platelet-rich plasma. Dermatol Surg. 2011 Apr;37(4):463-8. doi: 10.1111/j.1524-4725.2011.01916.x. PMID 21481064
- [Background] Hui Q, Chang P, Guo B, Zhang Y, Tao K. The Clinical Efficacy of Autologous Platelet-Rich Plasma Combined with Ultra-Pulsed Fractional CO2 Laser Therapy for Facial Rejuvenation. Rejuvenation Res. 2017 Feb;20(1):25-31. doi: 10.1089/rej.2016.1823. Epub 2016 Jun 23. PMID 27222038
- [Background] Kieb M, Sander F, Prinz C, Adam S, Mau-Moller A, Bader R, Peters K, Tischer T. Platelet-Rich Plasma Powder: A New Preparation Method for the Standardization of Growth Factor Concentrations. Am J Sports Med. 2017 Mar;45(4):954-960. doi: 10.1177/0363546516674475. Epub 2016 Dec 13. PMID 27903591
- [Background] Goodman GJ, Baron JA. Postacne scarring--a quantitative global scarring grading system. J Cosmet Dermatol. 2006 Mar;5(1):48-52. doi: 10.1111/j.1473-2165.2006.00222.x. PMID 17173571